CLINICAL TRIAL: NCT02756338
Title: BioMonitor 2 In-Office Setting Insertion Safety and Feasibility Evaluation With Device Functionality Assessment
Acronym: BioInsight
Status: Completed | Type: Observational
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BioInsight
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-09

CONDITIONS: Insertable Cardiac Monitor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: BioMonitor 2 Insertable Cardiac Monitor

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of performing the BioMonitor 2 insertion procedure in an office setting.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for continuous monitoring with an insertable cardiac monitor
* Willing to be implanted in an office setting with only local anesthetic available
* Able to understand the nature of the study and provide informed consent
* Able and willing to complete all routine follow-up visits at the study site for the expected 90-day follow-up
* Able and willing to use a CardioMessenger® capable of communicating with the BioMonitor 2
* Age greater than or equal to 18 years

At the time of insertion, the following pre-procedure criteria must be met for the subject to undergo insertion:

* Most recent INR value (within 7 days) is less than 3.5 if currently taking warfarin
* Absence of infection with no history of infection within the last 30 days

Exclusion Criteria:

* Compromised immune system or at high risk of developing an infection
* Abnormal thoracic anatomy or scar tissue at the implant site that may adversely impact the insertion procedure
* Enrolled in any investigational cardiac device trial
* Currently indicated for or implanted with a pacemaker, ICD device, or hemodynamic monitoring system
* Currently implanted with an ICM or ILR
* Life expectancy less than 6 months
* Patients reporting pregnancy at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects indicated for continuous arrhythmia monitoring who are willing to undergo the insertion procedure in an office setting
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2016-06; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Flint, Michigan
  - Saginaw, Michigan
  - St Louis, Missouri
  - Greenville, North Carolina
  - Columbus, Ohio
  - Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Awad K, Weiss R, Yunus A, Bittrick JM, Nekkanti R, Houmsse M, Okabe T, Adamson T, Miller C, Alawwa AK. BioMonitor 2 in-office setting insertion safety and feasibility evaluation with device functionality assessment: results from the prospective cohort BioInsight study. BMC Cardiovasc Disord. 2020 Apr 15;20(1):171. doi: 10.1186/s12872-020-01439-8. PMID 32293279

RESULTS

PARTICIPANT FLOW:
Groups:
- BioMonitor 2 In-Office Setting Insertion Group: Post-market Study: Collecting safety and feasibility of performing office based insertion of a market-released insertable cardiac monitor.
Period: Overall Study
Arm/Group | BioMonitor 2 In-Office Setting Insertion Group
Started | 77
Completed | 72
Not Completed | 5
Not completed — Withdrawn by Investigator | 1
Not completed — Device Replaced with Pacemaker | 4

BASELINE CHARACTERISTICS:
Arm/Group | BioMonitor 2 In-Office Setting Insertion Group
Number analyzed (Participants) | 77
Age, Customized [Mean (Standard Deviation); unit: years]
  Age at Enrollment | 62.1 (15.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 71
  Black or African American | 5
  Race Not Specified | 1
  Not Hispanic or Latino Ethnicity | 76
  Ethnicity Not Specified | 1
Height [Mean (Standard Deviation); unit: inches] | 67.8 (4.82)
Weight [Mean (Standard Deviation); unit: pounds] | 205.6 (47.93)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Insertion Procedure-related Adverse Event That Requires Additional Invasive Intervention to Resolve
Description: In order to be included in the primary objective analysis, insertion procedure-related adverse events must also include resolution by invasive action such as device removal, device replacement, surgical repositioning of the device, or another surgery preformed related to the device or primary insertion procedure.
Time Frame: Insertion through 90 days
Population: The evaluable subject population is the sum of total unique subjects who completed the 90-day follow-up and/or who experienced a primary objective adverse event.
Measure: Number; unit: participants with a Primary Objective AE
Arm/Group | BioMonitor 2 In-Office Setting Insertion Group
Number analyzed (Participants) | 72
participants with a Primary Objective AE | 0

2. Secondary Outcome: Number of Participants With Insertion Procedure-related Adverse Event Not Included in Primary Objective
Description: All insertion procedure-related adverse events not included in the Primary Objective
Time Frame: Insertion through 90 days
Population: The evaluable subject population is the sum of total unique subjects who completed the 90-day follow-up and/or who experienced a secondary objective adverse event.
Measure: Count of Participants; unit: Participants
Arm/Group | BioMonitor 2 In-Office Setting Insertion Group
Number analyzed (Participants) | 73
Participants | 2

3. Secondary Outcome: Characterization of Insertion Procedure: Device Orientation
Description: Position A includes orientations at 45 degrees relative to the sternum over the fourth intercostal space, position B includes orientations parallel to the sternum over the fourth intercostal space, and position C includes orientations perpendicular to the sternum and sub-mammary.
Time Frame: At insertion
Population: All subjects who underwent insertion
Measure: Count of Participants; unit: Participants
Arm/Group | BioMonitor 2 In-Office Setting Insertion Group
Number analyzed (Participants) | 77
Participants
  Position A | 35
  Position B | 38
  Position C | 1
  Other | 3

4. Secondary Outcome: Characterization of Insertion Procedure: Incision Size
Time Frame: At insertion
Population: Number of participants analyzed included all subjects with a reported incision size. Incision size was not collected or reported for 3 participants.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | BioMonitor 2 In-Office Setting Insertion Group
Number analyzed (Participants) | 74
millimeters | 14.9 (3.74)

5. Secondary Outcome: Characterization of Insertion Procedure: Procedure Duration
Time Frame: At insertion
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | BioMonitor 2 In-Office Setting Insertion Group
Number analyzed (Participants) | 77
minutes | 8.4 (3.69)

6. Secondary Outcome: Characterization of Device Functionality Post-insertion: R-wave Amplitudes
Description: This includes average R-wave amplitudes collected at insertion, wound check, and 90-day study visits. Long-term trends available through Home Monitoring from insertion through the 90-day study period was also collected and presented as a separate average.
Time Frame: Insertion, Wound Check (5 to 14 days post-insertion), 90-day (75 to 120 days post-insertion)
Population: Five subjects did not complete their 90-day visits as reported in Participant Flow and therefore data was not collected for those visits. Only one subject did not transmit to Home Monitoring due to poor reception and therefore there was no data for this patient in Home Monitoring.
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | BioMonitor 2 In-Office Setting Insertion Group
Number analyzed (Participants) | 77
millivolts (mV)
  Insertion Procedure Visit | 0.77 (0.5)
  Wound Check Visit | 0.69 (0.4)
  90-day Follow-up Visit: number analyzed (Participants) | 72
  90-day Follow-up Visit | 0.67 (0.3)
  Home Monitoring 90-day Average: number analyzed (Participants) | 76
  Home Monitoring 90-day Average | 0.68 (0.34)

ADVERSE EVENTS:
Time Frame: Insertion through 90 days
Arm/Group | BioMonitor 2 In-Office Setting Insertion Group
All-Cause Mortality (participants affected / at risk) | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77
Other Adverse Events (participants affected / at risk) | 2/77
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BioMonitor 2 In-Office Setting Insertion Group (N=77)
Secondary Infection (Surgical and medical procedures) | 1 (1)
Surrounding Tissue Damage (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators agree to submit copies of any manuscript proposed for publication to Sponsor for review at least 30 days in advance of submission for publication or presentation. Sponsor may extend such review period another 90 days to file patent applications to take other steps to protect its intellectual property interests, or to remove from the paper or presentation any language that is detrimental to Sponsor's intellectual property interests.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT02756338/Prot_SAP_000.pdf